CLINICAL TRIAL: NCT01560910
Title: Detection of Minimal Change Esophagitis by I-scan
Status: Completed | Type: Observational
Sponsor: arpa pungrasamee (Other)
Responsible Party: Sponsor-Investigator, arpa pungrasamee, Doctor, Maharaj Nakorn Chiang Mai Hospital
Organization: Maharaj Nakorn Chiang Mai Hospital (Other)
Other Study IDs: ISSNEXI0018
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Gastro-esophageal Reflux Disease; Non-erosive Reflux Disease
Keywords: with or without GERD symptoms; presenting to gastrointestinal clinic of Maharaj Nakorn Chiangmai Hospital; November 2009 to November 2010; GERD; NERD
MeSH Terms: conditions — Gastroesophageal Reflux; Non-Erosive Reflux Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study design and objective The primary outcome of this prospective cohort study was to identify the endoscopic findings that have diagnostic value for the prediction of NERD (minimal change esophagitis) by using HD endoscopy with i-scan. The secondary outcome was to evaluate the response to proton pump inhibitor (PPI) in GERD patients with or without minimal change esophagitis.

DETAILED DESCRIPTION:
Background and aims Majority of patients with gastro-esophageal reflux disease (GERD) were non-erosive reflux disease (NERD). High definition (HD) endoscopy with i-scan could enhance visualization of mucosal and vascular pattern and might identify changes that were invisible at standard endoscopy. This study aimed to evaluate the endoscopic findings that may have diagnostic value for the prediction of NERD by using HD endoscopy with i-scan.

Methods Patients with typical GERD symptoms and healthy control without GERD symptoms were included and 2 validated GERD questionnaires were completed. The endoscopist was blinded to the presence of reflux symptoms and distal esophagus was examined using standard white light endoscopy followed by i-scan. Mucosal morphology at squamocolumnar junction (SCJ) observed by i-scan were compared between GERD patients and controls.

ELIGIBILITY:
Inclusion Criteria:

18 to 80 years of age and had ability to provide written informed consent

Exclusion Criteria:

1. pregnancy,
2. cirrhosis or presence of gastroesophageal varices,
3. gastrointestinal hemorrhage,
4. angina pectoris,
5. allergy to PPI,
6. high risk or contraindication for endoscopy,
7. chronic cough,laryngitis, asthma.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients with or without GERD symptoms presenting to gastrointestinal clinic of Maharaj Nakorn Chiangmai Hospital from November 2009 to November 2010 were invited to participate in this study. All patients completed 2 validated questionnaires (RDQ: reflux diagnostic questionnaire and HRQL: Health-related quality-of-life GERD questionnaire) after giving written informed consent. Patients were enrolled if they were 18 to 80 years of age and had ability to provide written informed consent.
  Patients who have heartburn or regurgitation more than 2 times/week for at least 1 month were defined as having GERD and patient without any reflux symptoms served as controls.The exclusion criteria were 1) pregnancy, 2) cirrhosis or presence of gastroesophageal varices, 3) gastrointestinal hemorrhage, 4) angina pectoris, 5) allergy to PPI, 6) high risk or contraindication for endoscopy, 7) chronic cough, laryngitis, asthma.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Maharaj Nakorn Chiangmai Hospital, Chiang Mai, Thailand